CLINICAL TRIAL: NCT00080366
Title: Treatment Efficacy of 1-Octanol Compared to Placebo in Adults With Essential Tremor
Brief Title: Octanol to Treat Essential Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040147; 04-N-0147
Record Dates: First submitted 2004-03-27; First posted 2004-03-29 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-03

CONDITIONS: Essential Tremor
Keywords: Essential Tremor; Cross over Design; Accelerometry; Placebo; Alcohol Responsive; Double Blind; 1-Octanol
MeSH Terms: conditions — Essential Tremor | interventions — 1-Octanol

INTERVENTIONS:
Drug: 1-Octanol

SUMMARY:
This study will evaluate the effectiveness of 1-octanol, a substance similar to alcohol but less intoxicating, for treating essential tremor. Essential tremor is an involuntary shaking, usually of the hands, for which there is no satisfactory treatment. It affects about 1.4 percent of the general U.S. population, with the figure climbing to nearly 4 percent among people over 40. Results of two previous NIH studies have shown 1-octanol to be promising as a potential new treatment. This study will test the effectiveness of 1-octanol on essential tremor at doses lower than those given previously.

Patients 21 years old and older with essential tremor may be eligible for this study. Participants are admitted to the NIH Clinical Center for two treatment periods of 1 week each, with a 1-week break at home between treatments. Before beginning treatment, participants undergo a medical history, physical examination, blood and urine tests, and an electrocardiogram (EKG). In addition, tremors are measured using accelerometry, a procedure in which a small device, mounted on a piece of cardboard, is taped to the patient's hand for about 30 minutes.

Patients are randomly assigned to one of two groups. One group takes 2 to 4 capsules of 1-octanol 3 times a day for 1 week, followed by a 1-week "washout" period (no treatment), and then 2 to 4 capsules of placebo 3 times a day for 1 week. Following the same dosage schedule, the second group takes placebo the first week, followed by the washout period and then 1-octanol treatment. Blood pressure and pulse are measured at 15, 30, and 60 minutes after the first dose of the day and then 3 times a day each day of hospitalization, EKG and blood draws are done every other day during hospitalization, and blood is drawn again 1 week after the end of the study. Patients evaluate their tremor daily according to a tremor scale and are also rated according to an alcohol intoxication scale.

DETAILED DESCRIPTION:
Essential tremor is a very common movement disorder affecting approximately 1.4% of the population. Response to medications such as beta blockers and mysoline may be only partial or be accompanied by intolerable side effects. Roughly 80% of patients have significant tremor reduction from? ethanol although daily use of this as a treatment has potentially serious social and legal consequences. The leading hypothesis for the pathophysiology of essential tremor is the unmasking of spontaneous oscillation of neurons in the inferior olive. Both ethanol and 1-octanol have been shown to reduce these spontaneous oscillations in a animal model of essential tremor; however, 1-octanol does this at a dose much lower than an intoxicating dose suggesting that it may be useful in the treatment of essential tremor. Two pilot studies with 1-octanol in patients with essential tremor suggested it was both efficacious and safe.

Objectives: The aim of the present study is to further assess efficacy of 1-octanol in essential tremor in a double-blinded, placebo-controlled study.

Study population: Patients with alcohol-responsive essential tremor.

Design: Double-blind, placebo-controlled two-period cross-over design.

Outcome parameters: Primary outcome parameter is tremor as assessed by accelerometry, secondary outcome measures are spiral drawing, subjective and clinical scoring.

Estimate of the outcome: 1-octanol at the dose of 32mg/kg three times a day will significantly improve tremor in patients with alcohol-responsive essential tremor.

Anticipated risks and benefits: Besides the unusual taste, there are no anticipated risks associated with 1-octanol ingestion. Patients may experience an improvement of their tremor.

Potential meaning for the field: Better treatment of essential tremor.

ELIGIBILITY:
* INCLUSION CRITERIA:

  14 patients with a clinical diagnosis of essential tremor will participate in the study. Selection criterion is essential tremor with a history of ethanol responsiveness. Informed consent will be obtained by any of the co-investigators.

Patients must be off any medications used to treat essential tremor such as mysoline or propranolol for at least 2 weeks. Patients must withhold ethanol and caffeine 24 hours prior to starting the treatment periods through the end of treatment periods, including alcohol or caffeine containing over the counter medications. Ethanol and caffeine consumption is allowed in the washout period.

EXCLUSION CRITERIA:

Patients with abnormalities on neurologic exam other than tremor.

Patients with a history of chronic alcohol dependence.

Patients with chronic medical conditions such as renal failure, hepatic failure and chronic lung disease.

Patients on other medications that cannot be temporarily discontinued for the length of the study.

Patients, who, for moral or religious reasons, do not wish to take a potentially intoxicating drug.

Patients with abnormalities on their baseline screening laboratory tests.

Women who are pregnant or lactating.

Patients under the age of 21.

Asians and Pacific Islanders.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14
Dates: Start 2004-03; Study Completion 2007-03

PRIMARY OUTCOMES:
Tremor as assessed by accelerometry.

SECONDARY OUTCOMES:
Spiral drawing, subjective and clinical scoring.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bikson M, Ghai RS, Baraban SC, Durand DM. Modulation of burst frequency, duration, and amplitude in the zero-Ca(2+) model of epileptiform activity. J Neurophysiol. 1999 Nov;82(5):2262-70. doi: 10.1152/jn.1999.82.5.2262. PMID 10561404